CLINICAL TRIAL: NCT00301002
Title: A Pilot Open-Label Study to Evaluate the Safety and Observe the Effectiveness of 16 Weeks of Alefacept in Palmar Plantar Pustulosis (IST 92)
Brief Title: Study to Evaluate the Efficacy of Alefacept to Treat Palmar Plantar Pustulosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Guenther Dermatology Research Centre (Other)
Collaborators: Biogen (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IST 92
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2006-11-23 (Estimated); Status verified 2006-11

CONDITIONS: Psoriasis; Palmoplantaris Pustulosis; Pustular Psoriasis of Palms and Soles; Pustulosis Palmaris et Plantaris; Pustulosis of Palms and Soles
Keywords: safety; effectiveness; Alefacept; Palmar; Plantar; Pustulosis
MeSH Terms: conditions — Psoriasis | interventions — Alefacept

INTERVENTIONS:
Drug: Alefacept

SUMMARY:
The purpose of this study is to determine if Alefacept is effective in the treatment of palmar plantar pustulosis.

DETAILED DESCRIPTION:
Palmar plantar pustulosis is a chronic, disabling skin condition which is difficult to treat since it is often recalcitrant to current treatments and associated with high recurrence rates. This condition appears to be a T lymphocyte mediated condition and is thought by some to be a subtype of psoriasis. Alefacept affects T cell activation and induces apoptosis of memory T cells. It has been shown to be efficacious in the treatment of psoriasis vulgaris and may be associated with prolonged remissions. There is extremely limited experience with use of Alefacept in Palmar Plantar Pustulosis. This pilot trial should provide additional information concerning its use for this indication.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have stable, moderate, severe or very severe palmar plantar pustulosis.
* Must have a minimum of at least 3 pustules on 1 sole or palm.
* Must give written informed consent.
* Subjects must be 18 years of age or older.
* Adult Males and non-pregnant, non-lactating females.
* Female subjects of childbearing potential must state that they are using measures to avoid conception through active means.
* Subjects must be in general good health with no other skin disease, disease state or physical condition which would impair evaluation of palmar plantar pustulosis or which would increase their health risk by study participation.
* Subjects must be willing to receive a 15 mg IM injection of Alefacept weekly for 16 weeks.

Exclusion Criteria:

* Female subjects who are not postmenopausal for at least 1 year, surgically sterile, or willing to practice effective contraception during the study. Nursing mothers, pregnant women and women planning to become pregnant while on study are to be excluded.
* Current enrollment in any investigational study in which the subject is receiving any type of drug, biologic, or non-drug therapy.
* Serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., pneumonia, septicemia) within the 3 months prior to the first dose of investigational drug.
* Any subject whose CD4+ T-lymphocyte count at study entry is less than the lower limit of normal per reference laboratory.
* Treatment with another investigational drug or approved therapy for investigational use within 28 days prior to investigational drug administration.
* Treatment with psoralen + ultraviolet A (PUVA), systemic retinoids, systemic steroids, methotrexate, cyclosporine, azathioprine, thioguanine, etanercept, efalizumab, infliximab, adalimumab or mofetil or other systemic immunosuppressant agents within the 28 days prior to investigational drug administration.
* Ultraviolet B (UVB) phototherapy within 14 days prior to investigational drug administration.
* Treatment within 7 days with topical agents (e.g. tar, anthralin, calcipotriol, tazarotene, steroids) which might have an effect on palmar plantar pustulosis.
* Known HIV, Hepatitis B or C seropositivity or tuberculosis infection.
* Significant abnormal chemistry, i.e. liver function tests greater than 3 times the upper limit of normal.
* Allergy to Alefacept or any of the components of the formulation.
* Known malignancy or history of malignancy within the previous 5 years (with the exception of basal cell carcinoma of the skin or squamous cell carcinoma in situ of the skin that has been treated with no evidence of recurrence.)
* Previous treatment with alefacept.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2005-06; Study Completion 2006-10

PRIMARY OUTCOMES:
percentage change in PPPASI from baseline

SECONDARY OUTCOMES:
number of subjects with PPPASI 75
number of subjects with PPPASI 50
number of subjects with very mild/clear PGA
number of subjects with no pustules

CONTACTS AND LOCATIONS:
Overall Officials: Lyn C Guenther, MD, FRCPC, Principal Investigator — The Guenther Dermatology Research Centre
Locations (1):
- The Guenther Dermatology Research Centre, London, Ontario, Canada